CLINICAL TRIAL: NCT02203409
Title: Laparoscopic Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shuguo Zheng, MD (Other)
Responsible Party: Sponsor-Investigator, Shuguo Zheng, MD, Professor of Hepatobiliary Surgery Institute; Chief Physician; Administrator of laparoscopic department, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Other Study IDs: SWHZSG005; 30972948 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2014-07-23; First posted 2014-07-29 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Liver Tumor
Keywords: liver tumor; Two stage hepatectomy; Hypertrophy; laparoscopy; ALPPS
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypertrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Laparoscopic ALPPS group: Patients with small future liver remnant who are operated with the "Associating Liver Partition and Portal vein ligation for Staged hepatectomy" approach
  Interventions: Procedure: Laparoscopic ALPPS

INTERVENTIONS:
Procedure: Laparoscopic ALPPS — Laparoscopic Associating Liver Partition and Portal Vein Ligation for Two-stage Hepatectomy

SUMMARY:
The purpose of this research is evaluate the results with laparoscopic ALPPS procedure in a single center. The validity, feasibility and limitations were assessed objectively through our clinical prospective study.The investigators expect laparoscopic ALPPS is safe, effective and feasible.

DETAILED DESCRIPTION:
Background: Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS) is a breakthrough in the field of hepatobiliary surgery in recent years，which stimulates the remnant liver volume(RLV) grew by 74%-87.2% in 9 to 13 days。The published literature reported that the two stages of ALPPS are the conventional laparotomy surgery，Patients need to undergo the injury of two open operations in a short time. The incidence of postoperative complications and mortality rate is as high as 53% -73% and 12%-27%.The aim of this study was to evaluate the results with laparoscopic ALPPS procedure in a single center, with special emphasis in validity, feasibility and limitations.

Results:

Clinical data include: operation time, intraoperative blood loss, volume of blood transfusion, complications and mortality, postoperative liver function, long-term curative effect and survival time were collected and analysed.

Statistical method:groups t-test ，univariate/multivariate analysis, logistic regression analysis, mixed linear regression, Cox survival analysis ，Kaplan-Meier survival analysis，Log-rank survival curves were used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with marginally resectable or primarily non-resectable locally advanced liver tumors
* Insufficient future liver remnant (FLR) either in volume or quality

Exclusion Criteria:

* Unresectable liver metastases in the future liver remnant or unresectable extrahepatic metastases
* Severe portal hypertension
* High anesthesiological risk
* Unresectable primary tumor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Safety of the procedure defined as the incidence of postoperative complications and mortality | within the first 90 days after the first stage

SECONDARY OUTCOMES:
survival rate | 3 years
  follow-up after the surgery every 3months, to understand relapse, death, statistics 1-year, 3-year overall survival rates，disease-free survival rates , recurrence and metastasis rate.

CONTACTS AND LOCATIONS:
Overall Officials: Shuguo Zheng, Study Director — Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, China

REFERENCES:
- [Background] Gruttadauria S, Vasta F, Minervini MI, Piazza T, Arcadipane A, Marcos A, Gridelli B. Significance of the effective remnant liver volume in major hepatectomies. Am Surg. 2005 Mar;71(3):235-40. PMID 15869140
- [Background] Barbaro B, Caputo F, Tebala C, Di Stasi C, Vellone M, Giuliante F, Nuzzo G, Bonomo L. Preoperative right portal vein embolisation: indications and results. Radiol Med. 2009 Jun;114(4):553-70. doi: 10.1007/s11547-009-0383-9. Epub 2009 Apr 13. English, Italian. PMID 19367466
- [Background] de Baere T, Denys A, Madoff DC. Preoperative portal vein embolization: indications and technical considerations. Tech Vasc Interv Radiol. 2007 Mar;10(1):67-78. doi: 10.1053/j.tvir.2007.08.003. PMID 17980321
- [Background] Alvarez FA, Ardiles V, Sanchez Claria R, Pekolj J, de Santibanes E. Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS): tips and tricks. J Gastrointest Surg. 2013 Apr;17(4):814-21. doi: 10.1007/s11605-012-2092-2. Epub 2012 Nov 27. PMID 23188224
- [Background] Schnitzbauer AA, Lang SA, Goessmann H, Nadalin S, Baumgart J, Farkas SA, Fichtner-Feigl S, Lorf T, Goralcyk A, Horbelt R, Kroemer A, Loss M, Rummele P, Scherer MN, Padberg W, Konigsrainer A, Lang H, Obed A, Schlitt HJ. Right portal vein ligation combined with in situ splitting induces rapid left lateral liver lobe hypertrophy enabling 2-staged extended right hepatic resection in small-for-size settings. Ann Surg. 2012 Mar;255(3):405-14. doi: 10.1097/SLA.0b013e31824856f5. PMID 22330038
- [Background] Sala S, Ardiles V, Ulla M, Alvarez F, Pekolj J, de Santibanes E. Our initial experience with ALPPS technique: encouraging results. Updates Surg. 2012 Sep;64(3):167-72. doi: 10.1007/s13304-012-0175-y. Epub 2012 Aug 18. PMID 22903531
- [Background] Li J, Girotti P, Konigsrainer I, Ladurner R, Konigsrainer A, Nadalin S. ALPPS in right trisectionectomy: a safe procedure to avoid postoperative liver failure? J Gastrointest Surg. 2013 May;17(5):956-61. doi: 10.1007/s11605-012-2132-y. Epub 2013 Jan 4. PMID 23288719
- [Background] Dokmak S, Belghiti J. Which limits to the "ALPPS" approach? Ann Surg. 2012 Sep;256(3):e6; author reply e16-7. doi: 10.1097/SLA.0b013e318265fd64. No abstract available. PMID 22895355
- [Background] Toyosaka A, Okamoto E, Mitsunobu M, Oriyama T, Nakao N, Miura K. Intrahepatic metastases in hepatocellular carcinoma: evidence for spread via the portal vein as an efferent vessel. Am J Gastroenterol. 1996 Aug;91(8):1610-5. PMID 8759671 (Retraction: PMID 9517679 Am J Gastroenterol. 1998 Mar;93(3):492)
- [Background] Yin Z, Fan X, Ye H, Yin D, Wang J. Short- and long-term outcomes after laparoscopic and open hepatectomy for hepatocellular carcinoma: a global systematic review and meta-analysis. Ann Surg Oncol. 2013 Apr;20(4):1203-15. doi: 10.1245/s10434-012-2705-8. Epub 2012 Oct 26. PMID 23099728
- [Background] Poon RT, Fan ST, Lo CM, Ng IO, Liu CL, Lam CM, Wong J. Improving survival results after resection of hepatocellular carcinoma: a prospective study of 377 patients over 10 years. Ann Surg. 2001 Jul;234(1):63-70. doi: 10.1097/00000658-200107000-00010. PMID 11420484